CLINICAL TRIAL: NCT02457260
Title: Study of the Utility of Oral Nitrite Therapy to Improve Skeletal Muscle Bioenergetics and Physical Capacity in Older Heart Failure Patients
Brief Title: Oral Nitrite for Older Heart Failure Patients
Acronym: ONTx+HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gladwin, Mark, MD (Individual)
Responsible Party: Principal Investigator, Daniel Forman, MD, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO15020481
Record Dates: First submitted 2015-05-12; First posted 2015-05-29 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Sodium Nitrite

STUDY DESIGN:
Intervention Model Description: Healthy Controls vs Heart Failure with reduced Ejection Fraction (HFrEF) vs Heart Failure with preserved Ejection Fraction (HFpEF) on four weeks of nitrite treatment tid.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy control (Experimental): 10 healthy adults, age 70 or older to receive 14 Nitrogen (14N) sodium nitrite, 40 mg tid
  Interventions: Drug: 14 N Sodium Nitrite
- HFpEF (Experimental): 10 adults with heart failure and preserved ejection fraction age 70 or older to receive 14N sodium nitrite, 20 or 40 mg tid depending on dose stratification for safety
  Interventions: Drug: 14 N Sodium Nitrite
- HFrEF (Experimental): 10 adults with heart failure and reduced ejection fraction aged 70 or older to receive 14N sodium nitrite, 20 or 40 mg tid depending on dose stratification for safety
  Interventions: Drug: 14 N Sodium Nitrite

INTERVENTIONS:
Drug: 14 N Sodium Nitrite — oral formulation of sodium nitrite 40 mg three times daily for 4 weeks
  Other Names: sodium nitrite

SUMMARY:
Studies have demonstrated nitrite therapy increases adenosine triphosphate (ATP) synthesis in skeletal muscle mitochondria concomitant with reduced whole-body oxygen cost during steady state exercise. Our own work has demonstrated safety and efficacy of an FDA investigational new drug (IND) approved sodium nitrite (10 milligram [mg]) capsule, and its utility to upregulate the sirtuin 3 adenosine monophosphate protein kinase (SIRT3-AMP) pathway of skeletal muscle of younger heart failure (HF) patients. It now seems exceptionally logical and opportune to apply these insights to older HF patients and to delineate mechanisms of disease and aging that respond to nitrite therapy.

DETAILED DESCRIPTION:
Heart failure (HF) is epidemic with aging and prevalence of HF is steadily increasing as the population of older adults expands. Despite the fact that age always stands out as a leading risk factor for HF incidence as well as for poor HF prognosis, few HF trials focus specifically on aging physiology as a key determinant of the disease, and/or on the utility of targeting mechanisms associated with aging as beneficial therapeutic targets. Consistently, HF trials have tended to focus primarily on central mechanisms of cardiac pumping dysfunction despite the fact that HF-outcomes are strongly related to functional decrements that are largely mediated by peripheral manifestations of the disease, and which are particularly interrelated with aging physiology. HF-related skeletal muscle myopathy is a manifestation of HF that diminishes physical function, and which is likely exacerbated by sarcopenia, vascular stiffening, and other aspects of aging such that exercise intolerance is disproportionate among older HF populations as well as its insidious clinical implications. In a pilot investigation, the investigators will study older (age ≥70 years) adults, including patients with HF with reduced ejection fraction (HFrEF) and HF with preserved ejection fraction (HFpEF) and age-matched healthy controls, to study benefits of nitrite therapy (in addition to established standards of HF care) to improve physical function. In this pilot analysis the investigators will focus on the utility of daily nitrite supplements to moderate aerobic (maximal and submaximal) and strength (maximal, endurance, and power) indices as well as underlying skeletal muscle mechanisms (skeletal muscle mitochondrial performance, gene expression, and capillarity).

Atrophy of type 1 skeletal muscle myocytes is associated with HFrEF and HFpEF. Multiple studies of normal aging have also demonstrated typical atrophy of type 2 skeletal muscle fibers. Consistently, older adults are compromised by cumulative atrophy risks, with studies showing losses of lean body mass as well as intrinsic skeletal muscle weakening, increased interstitial fat, and increased inflammation, with associated functional decrements and fatigue. While aerobic and strength exercise training may be used to modify such HF-related muscle patterns, deconditioning remains pervasive among older HF patients, and efforts to promote exercise interventions are typically confounded by comorbidity (e.g. arthritis, peripheral arterial disease, diabetes, depression), geriatric syndromes (e.g., falls, frailty, incontinence, dementia, poor sleep, malnutrition, auditory and vision impairments), as well as pain, anxiety, and logistic limitations. Even major exercise-training trials that provided strong reinforcements to ensure requisite behavioral changes yielded only poor exercise adherence. There is high conceptual rationale for a therapy that intrinsically improves skeletal muscle performance in HF as a vital means to improve physical function and moderate effects of disease itself as well as to frailties and enfeeblement associated with the disease. This will potentially improve efficacy and quality of care, and also potentially mitigate the skyrocketing costs associated with aggregate HF management.

Studies have demonstrated nitrate therapy increases adenosine triphospate (ATP) synthesis in skeletal muscle mitochondria concomitant with reduced whole-body oxygen cost during steady state exercise. Our own work has demonstrated safety and efficacy of an FDA-IND approved sodium nitrite (10 mg) capsule, and its utility to upregulate the SIRT3-AMP pathway of skeletal muscle of younger HF patients. It now seems exceptionally logical and opportune to apply these insights to older HF patients and to delineate mechanisms of disease and aging that respond to nitrite therapy.

Overall aims:

1. To demonstrate that oral nitrite pills provide skeletal muscle physiological benefit in old HFrEF and HFpEF patients:

   * To show that oral supplements are manifest as increased plasma nitrite.
   * To show that increased plasma nitrite is associated with improved skeletal muscle (mitochondrial respirometry) and platelet (Seahorse XF) metabolism.
   * To demonstrate that improved metabolism is associated with shifts in skeletal muscle anabolic gene expression (Fibronectin type III domain-containing protein 5 [FNDC5], peroxisome proliferator-activated receptor-γ coactivator [PGC1α], Sirtuin 3) as well as reduced catabolic gene expression (ubiquitin, muscle RING-Finger Protein [MuRF], Atrogin1]) and inflammation (Tumor necrosis factor alpha [TNFα], Interleukin 1beta (IL-1β), Interleukin six (IL-6).
2. To demonstrate that improved skeletal physiology achieved using oral nitrate pills is associated with improved clinical indices in old HFrEF and HFpEF patients:

   * To show that oral nitrite supplements increase efficiency of work, i.e., reduced oxygen uptake (VO2) required for the same work intensity.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria HF Population

* New York Heart Association (NYHA) class II or III for the previous three months despite a minimum of 6 weeks of treatment. Echo criteria will be confirmed as part of the initial study assessment.
* Age ≥70 years
* HFrEF patients left ventricular ejection fraction (LVEF) ≤40%
* HFpEF patients LVEF>40%, may include E/E' >8, left atrial size>40 mL/m2
* Optimal therapy according to American Heart Association (AHA)/American College of Cardiology(ACC) and Heart Failure Society of America (HFSa) HFrEF guidelines, including treatment with angiotensin-converting enzyme inhibitor (ACEI) and beta-blocker therapy (for at least 6 weeks), or have documented reason for variation, including medication intolerance, contraindication, patient preference, or personal physician's judgment.
* Patients using aspirin (ASA) will be eligible, but asked to hold the medication for 48 hours prior to biopsy. This technique has previously been used with consistent safety. Patients will also be asked to avoid non-steroidal anti-inflammatory medications (NSAIDs) for 48 hours prior to the biopsy.
* Patients using anti-thrombin and anti-platelet therapy will plan to modify prior to muscle biopsies individually in coordination with the participant's primary cardiologist.

Inclusion Criteria Age-Matched Control Population

* Age ≥70 years
* Absence of any type of cardiovascular disease.
* Absence of diabetes or other chronic disease processes

Exclusion Criteria:

Exclusion Criteria for All participants

* Allergy to lidocaine
* Dementia
* End-stage malignancy
* Orthopedic exercise limitation
* Chronic use of oral corticosteroids or other medications that affect muscle function.
* Chronic ethyl alcohol (ETOH) or drug dependency.
* Any bleeding disorder that would contraindicate biopsy such as history of clinically significant bleeding diathesis (e.g., Hemophilia A or B, Von Willebrand's Disease or congenital Factor VII deficiency).
* Psychiatric hospitalization within the last 3 months

Exclusion Criteria HF Population

* Major cardiovascular event or procedure within the prior 6 weeks.
* HF secondary to significant uncorrected primary valvular disease (except mitral regurgitation secondary to left ventricular dysfunction). If valve replacement has been performed, patient may not be enrolled for 12 months after this procedure.
* Severe valvular heart disease
* Mechanical valve replacement requiring warfarin
* Currently taking clopidogrel for a recent stent placement and/or a complex atherosclerotic lesion such that holding clopidogrel creates disproportionate risk.
* ICD (Internal cardiodefibrillator) device with heart rate limits that prohibit exercise assessments. Referring physicians will be provided with an opportunity to reprogram devices so that patients can participate.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01-08; Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Forman, MD, Principal Investigator — University of Pittsburgh; Mark Gladwin, MD, Study Director — University of Pittsburgh
Locations (1):
- UPMC Montefiore Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Control: 12 healthy adults, age 70 or older to receive 14 Nitrogen (14N) sodium nitrite, 40 mg tid
  14 N Sodium Nitrite: oral formulation of sodium nitrite 40 mg three times daily for 4 weeks
- HFpEF: 7 adults with heart failure and preserved ejection fraction age 70 or older to receive 14N sodium nitrite, 20 or 40 mg tid depending on dose stratification for safety
  14 N Sodium Nitrite: oral formulation of sodium nitrite 40 mg three times daily for 4 weeks
- HFrEF: 2 adults with heart failure and reduced ejection fraction aged 70 or older to receive 14N sodium nitrite, 20 or 40 mg tid depending on dose stratification for safety
  14 N Sodium Nitrite: oral formulation of sodium nitrite 40 mg three times daily for 4 weeks
Period: Overall Study
Arm/Group | Healthy Control | HFpEF | HFrEF
Started | 12 | 7 | 2
Completed | 10 | 4 | 1
Not Completed | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Heart Failure With Preserved Ejection Fraction (HFpEF): 7 adults with heart failure and preserved ejection fraction age 70 or older to receive 14N sodium nitrite, 20 or 40 mg tid depending on dose stratification for safety
  14 N Sodium Nitrite: oral formulation of sodium nitrite 40 mg three times daily for 4 weeks
- Heart Failure With Reduced Ejection Fraction(HFrEF): 2 adults with heart failure and reduced ejection fraction aged 70 or older to receive 14N sodium nitrite, 20 or 40 mg tid depending on dose stratification for safety
  14 N Sodium Nitrite: oral formulation of sodium nitrite 40 mg three times daily for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Heart Failure With Preserved Ejection Fraction (HFpEF) | Heart Failure With Reduced Ejection Fraction(HFrEF) | Total
Number analyzed (Participants) | 12 | 7 | 2 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 12 | 7 | 2 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 0 | 10
  Male | 6 | 3 | 2 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 7 | 2 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 7 | 2 | 21

OUTCOME MEASURES:

1. Primary Outcome: Skeletal Muscle Bioenergetics- Polymerase Chain Reaction (PCR)
Description: Obtained via analysis of skeletal muscle biopsy of the vastus lateralis, Polymerase chain reaction (PCR) to assess pertinent gene expression within the pathways of ubiquitin [muscle ring finger protein 1 (MuRF), Atrogin1, Forkhead Box 03 (FoxO)], additionally Fibronectin type III domain-containing protein 5, the precursor of irisin (FNDC5), Peroxisome proliferator-activated receptor gamma co activator 1-alpha (PGC1α), and Sirtuin 3 were assessed.
Time Frame: Baseline; PRE and 4 weeks; POST
Population: Health Control- 2 and 1 HFrEF participants have missing data for the gene analysis due to muscle samples not providing a clean reference value for inclusion of data analysis.. 6 subjects withdrawn from the study.
Measure: Mean (Standard Deviation); unit: Relative Expression
Groups:
- HFpEF: 4 adults with heart failure and preserved ejection fraction age 70 or older to receive 14N sodium nitrite, 20 or 40 mg tid depending on dose stratification for safety
  14 N Sodium Nitrite: oral formulation of sodium nitrite 40 mg three times daily for 4 weeks
- HFrEF: 1 adults with heart failure and reduced ejection fraction aged 70 or older to receive 14N sodium nitrite, 20 or 40 mg tid depending on dose stratification for safety
  14 N Sodium Nitrite: oral formulation of sodium nitrite 40 mg three times daily for 4 weeks
Arm/Group | Healthy Control | HFpEF | HFrEF
Number analyzed (Participants) | 8 | 4 | 0
Relative Expression
  PCR -FNDC5 -PRE: number analyzed (Participants) | 6 | 4 | 0
  PCR -FNDC5 -PRE | 12.04 (0.45) | 11.91 (0.53) |
  PCR- FNDC5-POST: number analyzed (Participants) | 6 | 4 | 0
  PCR- FNDC5-POST | 11.79 (0.48) | 11.76 (0.34) |
  PCR- Sirtuin 3-PRE: number analyzed (Participants) | 6 | 4 | 0
  PCR- Sirtuin 3-PRE | 9.25 (0.23) | 9.12 (0.10) |
  PCR-Sirtuin 3-POST: number analyzed (Participants) | 6 | 4 | 0
  PCR-Sirtuin 3-POST | 9.10 (0.18) | 9.07 (0.14) |
  PCR-MuRF-PRE: number analyzed (Participants) | 6 | 4 | 0
  PCR-MuRF-PRE | 11.64 (0.25) | 11.90 (0.22) |
  PCR-MuRF-POST: number analyzed (Participants) | 6 | 4 | 0
  PCR-MuRF-POST | 11.46 (0.21) | 11.57 (0.46) |
  PCR-Atrogin1-PRE: number analyzed (Participants) | 6 | 4 | 0
  PCR-Atrogin1-PRE | 13.41 (0.13) | 13.55 (0.38) |
  PCR-Atrogin1-POST: number analyzed (Participants) | 6 | 4 | 0
  PCR-Atrogin1-POST | 13.30 (0.25) | 13.12 (0.48) |
  PCR- FoX O-PRE: number analyzed (Participants) | 6 | 4 | 0
  PCR- FoX O-PRE | 10.93 (0.27) | 10.95 (0.44) |
  PCR- FoX O-POST: number analyzed (Participants) | 6 | 4 | 0
  PCR- FoX O-POST | 10.74 (0.30) | 10.81 (0.61) |
  PCR- PGC1α-PRE: number analyzed (Participants) | 6 | 4 | 0
  PCR- PGC1α-PRE | 10.03 (0.14) | 10.06 (0.27) |
  PCR- PGC1α-POST: number analyzed (Participants) | 6 | 4 | 0
  PCR- PGC1α-POST | 9.96 (0.22) | 9.70 (0.48) |

2. Primary Outcome: Skeletal Muscle Bioenergetics - Mitochondrial Function
Description: Obtained via analysis of skeletal muscle biopsy of the vastus lateralis, Mitochondrial function was assessed using respirometry (State 3.12).
Time Frame: Baseline; PRE and 4 weeks; POST
Population: 2 Controls, 1 HFpEF and 1 HFrEF have no data for mitochondrial function due to no FCCP response or potential cytochrome c response. 6 subjects withdrawn from the study.
Measure: Mean (Standard Deviation); unit: nmol O / sec/ mg
Arm/Group | Healthy Control | HFpEF | HFrEF
Number analyzed (Participants) | 8 | 3 | 0
nmol O / sec/ mg
  Mitochondrial function- Fiber 1 State 3.12 PRE | 108.88 (51.69) | 122.99 (46.75) |
  Mitochondrial function- Fiber 1 State 3.12 POST | 123.59 (35.82) | 169.77 (69.33) |
  Mitochondrial function- Fiber 2 State 3.12 PRE | 122.84 (29.92) | 229.03 (82.63) |
  Mitochondrial function- Fiber 2 State 3.12 POST | 124.68 (70.04) | 120.44 (26.74) |

3. Secondary Outcome: Serology-platelet Bioenergetics
Description: Platelet bioenergetics (using Seahorse XF analysis), i.e., including glycolytic(OLIGO) as well as basal and maximal respiratory rates and extracellular acidification rate.
Time Frame: Baseline; PRE and 4 weeks; POST
Population: Patients that completed pre post testing in each of the three arms were include in analysis. 6 subjects withdrawn from the study.
Measure: Mean (Standard Deviation); unit: pmol/minute
Arm/Group | Healthy Control | HFpEF | HFrEF
Number analyzed (Participants) | 10 | 4 | 1
pmol/minute
  Basal respiratory rates-PRE | 122.77 (35.21) | 110.17 (22.89) | 148.71 (0)
  Basal respiratory rates-POST | 120.44 (31.05) | 120.90 (29.67) | 119.78 (0)
  OLIGO OCR- PRE | 29.38 (14.05) | 34.59 (22.80) | 29.49 (0)
  OLIGO OCR- POST | 27.28 (8.15) | 29.81 (11.30) | 11.25 (0)
  maximal respiratory rates- PRE | 181.08 (56.28) | 157.00 (46.64) | 188.09 (0)
  maximal respiratory rates- POST | 185.52 (52.83) | 144.99 (50.01) | 89.31 (0)

4. Secondary Outcome: Measures of Physical Function- Cardiopulmonary Exercise Test (CPX)
Description: Continuous metabolic gas collection or a cardiopulmonary exercise test occurred during a constant speed-steady state treadmill walking protocol (1.5mph at a 0% grade) for 5 minutes. During the final minute of the walking protocol oxygen consumption (VO2) was assessed to determined if the patient reached steady state VO2. Steady state VO2 was assessed by a less than 5% change in VO2 for a 30 second period of time. The 30 second average time is represented below in units of measure ml/kg/min. This is to show change in efficiency of performance of the constant speed test a decrease in VO2 from pre to post indicates greater efficiency.
Time Frame: Baseline; PRE and 4 weeks; POST
Population: All patients that have both pre and post data were assessed for all three groups. 6 subjects withdrawn from the study.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Healthy Control | HFpEF | HFrEF
Number analyzed (Participants) | 9 | 4 | 1
ml/kg/min
  Pre | 13.29 (4.14) | 11.55 (0.66) | 10.05 (0)
  Post | 11.27 (2.76) | 11.79 (2.75) | 10.50 (0)

5. Secondary Outcome: Measures of Physical Function- Gait Speed
Description: 4 meter gait speed assessed as part of the short performance physical battery (SPPB). This assessment evaluates how long it take a person can cover four meters at their usual walking speed from a stop when a person says go. This was completed twice to find the fastest speed was used as the variable.
Time Frame: Baseline; PRE and 4 weeks; POST
Population: All patients that have both pre and post data were assessed for all three groups. 6 subjects withdrawn from the study.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Healthy Control | HFpEF | HFrEF
Number analyzed (Participants) | 10 | 4 | 1
seconds
  Gait Speed- Pre | 4.32 (0.78) | 5.6 (2.24) | 4.22 (0)
  Gait Speed- Post | 4.36 (0.74) | 5.36 (1.81) | 4.06 (0)

6. Secondary Outcome: Measures of Physical Function- Handgrip
Description: Handgrip is used as a measure of upper body strength. three trials on each hand were completed with the patient seated and the arm at a right angle. For the purposes of this analysis all trials were averaged together.
Time Frame: Baseline; PRE and 4 weeks; POST
Population: All patients that have both pre and post data were assessed for all three groups. 6 subjects withdrawn from the study.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Healthy Control | HFpEF | HFrEF
Number analyzed (Participants) | 10 | 4 | 1
kg
  Handgrip- PRE | 26.53 (7.69) | 27.02 (5.15) | 25.25 (0)
  Handgrip-POST | 26.5 (8.61) | 26.02 (4.23) | 25.41 (0)

7. Secondary Outcome: Measures of Physical Function- Balance
Description: Balance was assessed as part of the short performance physical battery (SPPB). This assessment evaluates three components of static stand (stands with their feet together), semi tandem (stand with the heal of one foot beside the toe of the other foot), Tandem (stands with one foot directly in front of the other). Each test is held for as many seconds as they can up to ten seconds. Static and semi tandem if held for 10 second counts as 1 point if not held it is 0 points, tandem stand if held for 10 second is 2 points, if held for 3 to9.99 it is 1 point, otherwise 0 points. Total points are added up for all balance tests for a composite score with the higher the score the better and maximum being 4, minimum 0.
Time Frame: Baseline; PRE and 4 weeks; POST
Population: All patients that have both pre and post data were assessed for all three groups. 6 subjects withdrawn from the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Control | HFpEF | HFrEF
Number analyzed (Participants) | 10 | 4 | 1
score on a scale
  SPPB (Balance) - PRE | 3.5 (0.71) | 3.25 (1.5) | 1 (0)
  SPPB (Balance)-POST | 3.4 (0.52) | 3.75 (0.5) | 3 (0)

8. Secondary Outcome: Quality of Life Assessment- In Heart Failure
Description: Kansas City Cardiomyopathy Questionnaire (KCCQ)- is a standard tool to assess the quality of life of the heart failure patients. An overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains with the higher the score (0-100) the better the health status.
Time Frame: Baseline; PRE and 4 weeks; POST
Population: Kansas City Cardiomyopathy Questionnaire (KCCQ)- is a standard tool to assess the quality of life of the heart failure patients. Control patients were not assessed via KCCQ given it is not a valid tool for healthy. All HF patients that completed pre and post assessment were analyzed. 6 subjects withdrawn from the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Healthy Control: 0 healthy adults, age 70 or older to receive 14 Nitrogen (14N) sodium nitrite, 40 mg tid
  14 N Sodium Nitrite: oral formulation of sodium nitrite 40 mg three times daily for 4 weeks
Arm/Group | Healthy Control | HFpEF | HFrEF
Number analyzed (Participants) | 0 | 4 | 1
scores on a scale
  KCCQ- PRE |  | 83.40 (13.54) | 94.79 (0)
  KCCQ-POST |  | 86.13 (18.04) | 84.90 (0)

9. Secondary Outcome: Serology-Inflammatory Marker
Description: Inflammatory marker (C-reactive protein [CRP])
Time Frame: Baseline; PRE and 4 weeks; POST
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Healthy Control | HFpEF | HFrEF
Number analyzed (Participants) | 10 | 4 | 1
mg/L
  CRP-PRE | 1.37 (1.4) | 0.58 (0.52) | 27.57 (0)
  CRP-POST | 0.97 (0.91) | 1.26 (1.14) | 5.43 (0)

10. Secondary Outcome: Serology-plasma Nitrite and Nitrate
Description: plasma nitrite and plasma nitrate levels pre and post 4 week intervention
Time Frame: Baseline; PRE and 4 weeks; POST
Population: On analysis of data for this report it was found that three control samples had been missed on initial running of nitrate/nitrite bring the N=7 for that assessment. 6 subjects withdrawn from the study.
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Healthy Control | HFpEF | HFrEF
Number analyzed (Participants) | 7 | 4 | 1
µm
  Plasma Nitrite- PRE | 2.43 (2.96) | 0.11 (0.04) | 0.04 (0)
  Plasma Nitrite- POST | 0.50 (0.33) | 0.35 (0.15) | 0.11 (0)
  Plasma Nitrate- PRE | 61.01 (15.64) | 34.91 (10.44) | 39.81 (0)
  Plasma Nitrate- POST | 75.30 (15.64) | 44.2 (5.97) | 67.68 (0)

11. Secondary Outcome: Serology-platelet Bioenergetics-1
Description: Platelet bioenergetics (using Seahorse XF analysis), i.e., extracellular acidification rate.
Time Frame: Baseline; PRE and 4 weeks; POST
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mpH/min
Arm/Group | Healthy Control | HFpEF | HFrEF
Number analyzed (Participants) | 10 | 4 | 1
mpH/min
  extracellular acidification rate -PRE | 3.78 (3.06) | 3.22 (3.02) | 7.34 (0)
  extracellular acidification rate -POST | 3.67 (2.61) | 3.96 (3.68) | 0.66 (0)

ADVERSE EVENTS:
Time Frame: patients were assessed over 4 weeks of the nitrite intervention
Arm/Group | Healthy Control | HFpEF | HFrEF
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 10/12 | 6/7 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Control (N=12) | HFpEF (N=7) | HFrEF (N=2)
Belly Pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 5 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 5 | 1
Impaired Depth Perception (Nervous system disorders) | 1 | 0 | 0
Knee Strain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
leg cramps (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
leg twinge (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lightheadedness (General disorders) | 3 | 0 | 1
Lumbrosacral strain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Malaise With Flu (Infections and infestations) | 2 | 0 | 0
Muscle tightness- upper leg (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
nausea (Infections and infestations) | 2 | 0 | 0
Nocturia (Renal and urinary disorders) | 3 | 0 | 0
Tension in Head (General disorders) | 1 | 0 | 0
URI (Renal and urinary disorders) | 2 | 0 | 0
Vomiting (General disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Cramp (General disorders) | 1 | 0 | 0
Twinge (General disorders) | 1 | 0 | 0
dizzy (General disorders) | 1 | 0 | 0
Itchy Eyes (General disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Blood Blister (General disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Insomnia (General disorders) | 0 | 1 | 0
Increase in poor coordination (General disorders) | 0 | 1 | 0
Scaly itchy patch on thigh (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
increased heart rate (Cardiac disorders) | 0 | 1 | 0
syncopal episode (Nervous system disorders) | 0 | 1 | 0
Chest tightness (Cardiac disorders) | 0 | 1 | 0
Change in blood pressure (Cardiac disorders) | 0 | 1 | 0
back pain resolved (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
leg cramps resolved (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Diastolic (Cardiac disorders) | 0 | 1 | 0
Shin spasm pain recurring (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT02457260/Prot_SAP_000.pdf